CLINICAL TRIAL: NCT04701567
Title: Diagnostik Und Evaluierung Hepato-pankreatiko-biliärer Erkrankungen Mittels Morphologischer Und Funktioneller Magnetresonanztomographie
Brief Title: Diagnostic and Evaluation of Hepato-pancreatico-biliary Disease With MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Caecilia Reiner, Staff Radiologist, University of Zurich
Other Study IDs: BASEC ID 2020-01313
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Liver Diseases; Pancreas Disease
MeSH Terms: conditions — Liver Diseases; Pancreatic Diseases | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Liver disease
  Interventions: Diagnostic Test: Magnetic resonance imaging
- Pancreatic disease
  Interventions: Diagnostic Test: Magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: Magnetic resonance imaging — Advanced multiparametric MRI techniques to diagnose hepatic and pancreatic disease

SUMMARY:
This is a retrospective review of images from patient data. There is no recruitment necessary for this study.

Research Question: Can advanced multiparametric MRI techniques improve the detection and characterization of focal and diffuse liver disease, accurately assess treatment response and predict patient outcomes based on longitudinal monitoring? Hypotheses: Advanced multiparametric MRI techniques improve the detection, characterization and response assessment of focal and diffuse liver disease and can predict serious liver related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspicion for or diagnosed focal and/or diffuse liver or pancreatic disease who underwent MRI of the abdomen.
* 18 years of age and older.

Exclusion Criteria:

* Age less than 18 years.
* Lack of MRI of the abdomen.
* Inadequate image quality.
* Documented rejection to participate in research studies

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion for or diagnosed focal and/or diffuse liver or pancreatic disease who underwent MRI of the abdomen.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathology findings in focal and/or diffuse liver disease | 1 year
  Pathology findings in focal and/or diffuse liver disease
Pathology findings in focal and/or diffuse pancreatic disease | 1 year
  Pathology findings in focal and/or diffuse pancreatic disease

CONTACTS AND LOCATIONS:
Overall Officials: Caecilia Reiner, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No